CLINICAL TRIAL: NCT02108873
Title: Factors Associated With Nonattendance at Scheduled Outpatient Appointments in a University General Hospital
Acronym: AU1
Status: Completed | Type: Observational
Sponsor: Hospital Italiano de Buenos Aires (Other)
Responsible Party: Principal Investigator, Diego Hernan Giunta, MD, MD, Hospital Italiano de Buenos Aires
Other Study IDs: 2262
Record Dates: First submitted 2014-04-06; First posted 2014-04-09 (Estimated); Last update posted 2015-03-24 (Estimated); Status verified 2015-03

CONDITIONS: Appointments and Schedules; Outpatient Clinics, Hospital/Economics
Keywords: Appointments and Schedules; Outpatient Clinics, Hospital/economics

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Retrospective Cohort: Adult patients who had scheduled an appointment for outpatient primary care. Patients were divided into two groups, including those who attended their scheduled appointment and those who missed it.

SUMMARY:
Our objectives were to estimate the prevalence of nonattendance at outpatient offices, to identify the characteristics of appointments for which nonattendance was more likely to occur, and to generate a predictive model that could be applied to each appointment to estimate the probability of nonattendance.

DETAILED DESCRIPTION:
Nonattendance at scheduled appointments at outpatient clinics is a common problem in general medical practice, representing a significant cost to the health care system, and resulting in disruption of daily work planning.Nonattendance at medical appointments has consequences not only for doctors (as it requires a greater use of resources and time), but also for patients, because there may be deterioration in the quality of care, and dissatisfaction associated with delays in obtaining a new appointment.

Previous studies have reported that nonattendance at scheduled appointments is most frequently associated with those patients attending follow-up appointments, generally those assigned to another professional, those with appointments on Fridays, and those with appointments assigned 1 - 2 weeks in advance. Nonattendance was also associated with younger patient age, greater psychological problems, and lower socioeconomic status.Furthermore, in patients with chronic diseases, the nonattendance rate was also reported to be lower. Clinical patient characteristics can be important predictors of nonattendance, but they required high quality electronic health records to predict nonattendance accurately In the United States and Europe, the nonattendance rate is estimated to be between 6.5%-55%; there is little evidence regarding nonattendance in Latin America. Many studies have described the prevalence and impact of nonattendance at scheduled medical appointments, and possible strategies to decrease the nonattendance rate. However, few studies have utilized the characteristics associated with nonattendance for building predictive models, which might better identify those patients who may not attend a scheduled appointment

ELIGIBILITY:
Inclusion Criteria:

* Over 17 years.
* Adults who attended, did not attend and cancelled a scheduled appointment at the Outpatient care system at the Italian Hospital of Buenos Aires (HIBA)

Exclusion Criteria:

* The refusal to register or to the informed consent process.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: We included all requested appointments (random consecutive sampling) between 2012 and 2013 (24 month). The sample was randomized to allocate a generation cohort (two-thirds of the sample) and a validation cohort (one third of the sample).
Sampling Method: Probability Sample
Enrollment: 10000 (Actual)
Dates: Start 2014-05; Primary Completion 2014-09 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Prevalence of non attendance, attendance and cancellation | Cohort study of 24 month
  Characterize, describe and compare the clinical and administrative characteristics of outpatients who didn't attend, attended and cancelled an appointment in internal medicine/primary health care, clinical subspecialties and surgical specialties.

SECONDARY OUTCOMES:
Clinical and administrative characteristics | Cohort study of 24 month
  Characterize, describe and compare the clinical and administrative characteristics of outpatients who didn't attend, attended and cancelled an appointment in internal medicine/primary health care, clinical subspecialties and surgical specialties.

CONTACTS AND LOCATIONS:
Overall Officials: Diego H Giunta, MD, Principal Investigator — Hospital Italiano de Buenos Aires
Locations (1):
- Hospital Italiano de Buenos Aires, Capital Federal, Buenos Aires, Argentina